CLINICAL TRIAL: NCT00828425
Title: Management of Diabetes Mellitus Patients With Retinopathy
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr. Med. Dirk Schneider - Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CCH-DUM-2008/1
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Retinopathy; Diabetes Mellitus
Keywords: Diabetes Mellitus; retinopathy; Management of diabetic patients with retinopathy
MeSH Terms: conditions — Retinal Diseases; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Diabetic patients with retinopathy

SUMMARY:
Aim of this NIS is to retrospectively document the management of diabetic patients with retinopathy in a naturalistic setting in Switzerland. Following elements are going to be analyzed:

* which medication are used to keep blood pressure under control?
* which medication are used for metabolic control?
* the average control level of metabolism and blood pressure is compliant with the international guidelines?
* laser photocoagulation plays a role in the control of metabolism and blood pressure?
* there are differences in the control of metabolism and blood pressure between patients with DM I or DM II?
* there is an influence of renal failure on the choose of medication?

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients
* Diabetic retinopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetic patients with diabetic retinopathy
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2008-12; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Blood lipids, glycemia, HbA1C, blood creatinine, proteinuria, body weight | every 3 months
evolution of diabetic retinopathy | every 3 months

SECONDARY OUTCOMES:
concomitant medication | every 3 months

CONTACTS AND LOCATIONS:
Locations (62):
- Switzerland (62):
  - Research Site, Diegten, Basel-Landschaft
  - Research Site, Laufen, Basel-Landschaft
  - Research Site, Dättwil, Canton of Aargau
  - Research Site, Hausen B. Brugg, Canton of Aargau
  - Research Site, Lenzburg, Canton of Aargau
  - Research Site, Lupfig, Canton of Aargau
  - Research Site, Muri, Canton of Aargau
  - Research Site, Rheinfelden, Canton of Aargau
  - Research Site, Schinznach Dorf, Canton of Aargau
  - Research Site, Spreitenbach, Canton of Aargau
  - Research Site, Basel, Canton of Basel-City
  - Research Site, Bern, Canton of Bern
  - Research Site, Moutier, Canton of Bern
  - Research Site, Unterseen, Canton of Bern
  - Research Site, Estavayer-le-Lac, Canton of Fribourg
  - Research Site, Fribourg, Canton of Fribourg
  - Research Site, Collonge-Bellerive, Canton of Geneva
  - Research Site, Geneva, Canton of Geneva
  - Research Site, Le Grand-Saconnex, Canton of Geneva
  - Research Site, Les Acacias, Canton of Geneva
  - Research Site, Versoix, Canton of Geneva
  - Research Site, Alle, Canton of Jura
  - Research Site, Lucerne, Canton of Lucerne
  - Research Site, Rothenburg, Canton of Lucerne
  - Research Site, Le Locle, Canton of Neuchâtel
  - Research Site, Kerns, Canton of Obwalden
  - Research Site, Schaffhausen, Canton of Schaffhausen
  - Research Site, Küssnacht, Canton of Schwyz
  - Research Site, Tuggen, Canton of Schwyz
  - Research Site, Oberuzwil, Canton of St. Gallen
  - Research Site, Rorschach, Canton of St. Gallen
  - Research Site, Sankt Gallen, Canton of St. Gallen
  - Research Site, Wangs, Canton of St. Gallen
  - Research Site, Aigle, Canton of Vaud
  - Research Site, Bassins, Canton of Vaud
  - Research Site, Bex, Canton of Vaud
  - Research Site, Chateau-d'Oex, Canton of Vaud
  - Research Site, Clarens, Canton of Vaud
  - Research Site, Eysins, Canton of Vaud
  - Research Site, Lausanne, Canton of Vaud
  - Research Site, Nyon, Canton of Vaud
  - Research Site, Prilly, Canton of Vaud
  - Research Site, Renens VD, Canton of Vaud
  - Research Site, Salavaux, Canton of Vaud
  - Research Site, St-Legier, Canton of Vaud
  - Research Site, Vevey, Canton of Vaud
  - Research Site, Bassersdorf, Canton of Zurich
  - Research Site, Egg, Canton of Zurich
  - Research Site, Winterthur, Canton of Zurich
  - Research Site, Ascona, Canton Ticino
  - Research Site, Locarno, Canton Ticino
  - Research Site, Lugano, Canton Ticino
  - Research Site, Viganello, Canton Ticino
  - Research Site, Chur, Kanton Graubünden
  - Research Site, Ilanz, Kanton Graubünden
  - Research Site, Samedan, Kanton Graubünden
  - Research Site, Kreuzlingen, Thurgau
  - Research Site, Ardon, Valais
  - Research Site, Evionnaz, Valais
  - Research Site, Savièse, Valais
  - Research Site, Sierre, Valais
  - Research Site, Sion, Valais